CLINICAL TRIAL: NCT03924700
Title: Outcomes Following Lumbar Discectomy Surgery in Lumbar Herniated Intervertebral Disc With Biportal Endoscopy Versus Open Microdiscectomy Technique: A Prospective, Multicenter, Single-blinded, Randomized Controlled Non-inferiority Trial
Brief Title: Biportal Endoscopic Discectomy Versus Microdiscectomy: RCT, Non-inferiority Trial
Acronym: BESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BESS_002
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Lumbar Herniated Intervertebral Disc
Keywords: Herniated intervertebral disc; Discectomy; Microscope; Biportal endoscopy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biportal endoscopic discectomy (Experimental): Biportal endoscopic discectomy for lumbar herniated intervertebral disc
  Interventions: Procedure: Biportal endoscopy
- Microdiscectomy (Active Comparator): Microdiscectomy for lumbar herniated intervertebral disc
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: Biportal endoscopy — Biportal endoscopic spine surgery (BESS)
  Arms: Biportal endoscopic discectomy
Procedure: Microdiscectomy — Using microscope for discectomy
  Arms: Microdiscectomy

SUMMARY:
This study is to compare the clinical outcome between the biportal endoscopic discectomy and microdiscectomy in herniated intervertebral disc of lumbar spine

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20 and 80
* patients who has radiating pain (VAS >=40) on lower extremities with HIVD
* patients who required one-level discectomy between L1 and S1
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form

Exclusion Criteria:

* Revision surgery
* Over spondylolisthesis Gr II
* Degenerative lumbar scoliosis (Cobb angle >20)
* patients with a history of other spinal diseases (compression fracture, spondylitis, tumor)
* women with positive pregnancy tests before the trial or who planned to become pregnant within the following 3 years
* patients with a history of malignant tumor or malignant diseases (but the cases of cured disease with no relapse for the past 5 years were included in the present study)
* patients with mental retardation or whose parents or legal guardians were older or had mental disabilities
* other patients viewed as inappropriate by the staff

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index (ODI) | at 1 year after surgery
  The ODI is based on a self-administered questionnaire measuring ''back-specific function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale. The ODI scores ranges from 0 to 100, with higher scores indicating severe symptoms.
  This is assessed by ODI survey at 1 year after surgery

SECONDARY OUTCOMES:
Change from baseline Oswestry disability index (ODI) | 3, 6, and 12, months, and every year, up to 5 year after operation
  The ODI is based on a self-administered questionnaire measuring ''back-specific function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale. The ODI scores ranges from 0 to 100, with higher scores indicating severe symptoms.
Change from baseline Visual Analog Pain Scale (VAS) | 4, 8, 12, 24, 48 hours, 2 weeks, 3, 6, and 12, months, and every year, up to 5 year after operation
  VAS is a measurement score that indicates pain severity status. VAS score comprised a 10-cm line with ''none'' (0) on one end of the scale and ''disabling pain'' (10) on the other.
Change from baseline EuroQoL-5 dimension (EQ-5D) value | 3, 6, and 12, months, and every year, up to 5 year after operation
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Rated level can be coded as a number 1 to 5, which indicates having no problems for 1, and having extreme problems for 5. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 55555 (having extreme problems in all dimensions). EQ-5D health states may be converted into a single index value. The index values are a major feature of the EQ-5D instrument, facilitating the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions. The value sets are anchored on 11111 = 1 and 55555 = 0 and can therefore be used in QALY calculations.
Change from baseline PainDETECT score | 3, 6, and 12, months, and every year, up to 5 year after operation
  The painDETECT Questionnaire (PDQ) is a screening tool designed to detect neuropathic pain in patients with chronic low back pain (LBP) based on self-reported pain characteristics. The degree of the seven types of pain quality, the type of pain pattern, and the presence of radiating pain. From the three components of the PDQ, a total score is calculated; a high score indicates that the pain is likely to have a neuropathic component. Scoring is performed using a scoring manual, and results in a final screening score: a score of 0-12 indicates nociceptive pain, 19-38 indicates neuropathic pain, and 13-18 indicates mixed pain.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 1 month after operation
  Surgery related adverse events (incidental durotomy, wound infection, re-operation, re-admission)
Operation duration time (minutes) | Immediate after operation
  Intraoperative time in minutes
Volume of postoperative drainage (ml) | Within 3 days after operation
  Total drainage after surgery in milli-liter
Number of participants with complete discectomy | Within 3 days after operation
  After surgery, degree of discectomy was measured using postoperative MRI
Concentration of creatine phosphokinase level in blood | At 2 day after surgery
  Creatine phosphokinase assessment to measure muscle injury at operation
Volume of postoperative Fentanyl consumption | At 3 days after operation
  Total amount of fentanyl consumption after surgery (PCA dose + rescue dose)
Times of hospital stay (hours) | Within 7 days after operation
  Total hospital stay after surgery
Number of radiographic complications | every year, up to 5 year after operation
  Radiographic complications includes disc degeneration, facet degeneration, re-ruptured disc, back muscle atrophy, kyphotic change, disc rupture...

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyounggido
  - Chungnam National University Hospital, Daejeon